CLINICAL TRIAL: NCT00399763
Title: A Randomized, Placebo-controlled Trial of Atomoxetine for Attention Deficit Hyperactivity Disorder in Adolescents With Substance Use Disorder (SUD)
Brief Title: Atomoxetine for Attention Deficit Hyperactivity Disorder in Adolescents With Substance Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-0563
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; Substance Abuse
Keywords: Adolescent; ADHD; SUD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Substance-Related Disorders | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo plus individual cognitive behavioral therapy
  Interventions: Drug: Placebo
- 2 (Experimental): atomoxetine plus individual cognitive behavioral therapy
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Half of participants are randomized to atomoxetine plus individual cognitive behavioral therapy targeting substance use disorder
  Other Names: Strattera
  Arms: 2
Drug: Placebo — Half of participants are randomized to placebo plus individual cognitive behavioral therapy targeting substance use disorder
  Arms: 1

SUMMARY:
The purpose of this study is to find out whether atomoxetine (also called Strattera) helps teenagers (12-19) with Attention Deficit Hyperactivity Disorder (ADHD) and drug/alcohol problems.

DETAILED DESCRIPTION:
Evidence-based psychosocial treatments have recently been developed. However, very little data exist on the use of pharmacotherapy for adolescents SUD (Substance Use Disorder). One promising pharmacotherapy approach is to treat co-occuring psychiatric disorders. A common co-occurring disorder in adolescent SUD is attention-deficit/hyperactivity disorder (ADHD). Fortunately, new ADHD medications, such as atomoxetine, that do not have addictive potential are now available. However, all controlled studies of atomoxetine have specifically excluded teens with SUD. Therefore, little data exist on the safety and efficacy of the medication in this population. This research project will address the important research gap with the specific aim: to conduct a randomized, placebo-controlled trial of atomoxetine for ADHD in teens with SUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-19
* Provided assent/consent
* attention-deficit hyperactivity disorder (ADHD) by Kiddie Schedule for Affective Disorders and Schizophrenia (KSADS)
* Diagnostic and statistical manual of mental disorders, 4th edition (DSM-IV) checklist <=22
* At least one non-nicotine substance use disorder (SUD) by KSADS
* Plans to live locally for 4 months
* Willing to participate in cognitive behavioral therapy (CBT)

Exclusion Criteria:

* No mental illness that cannot be managed as an outpatient or without concurrent psychotropic medication
* No allergy to atomoxetine
* No narrow angle glaucoma
* No serious medical illness
* Not pregnant
* Not unwilling to use an effective form of contraception during the trial
* No SUD that cannot be managed as an outpatient or without concurrent psychotropic medication

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2005-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Thurstone, MD, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Thurstone C, Riggs PD, Salomonsen-Sautel S, Mikulich-Gilbertson SK. Randomized, controlled trial of atomoxetine for attention-deficit/hyperactivity disorder in adolescents with substance use disorder. J Am Acad Child Adolesc Psychiatry. 2010 Jun;49(6):573-82. doi: 10.1016/j.jaac.2010.02.013. PMID 20494267

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: The participants received placebo plus CBT for their substance use disorder for 12 weeks.
- Atomoxetine: The participants received atomoxetine for their ADHD and CBT for their substance use disorder. The atomoxetine was titrated to 100 mg daily unless participants were less then 70 kg. In that case, they were titrated to 1.2 mg/kg per day.
Period: Overall Study
Arm/Group | Placebo | Atomoxetine
Started | 35 | 35
Completed | 33 | 32
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Atomoxetine | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31 | 33 | 64
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.11 (1.78) | 16.06 (1.35) | 16.09 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 15
  Male | 30 | 25 | 55
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Change in Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) Attention-deficit/Hyperactivity Disorder (ADHD) Checklist
Description: All 18 ADHD symptoms are rated on a scale of 0 (none) to 3 (severe) since the previous study visit. The scores are summed to create a total ADHD severity scale score ranging from 0 (none) to 54 (most severe). A single value of mean change in ADHD severity for each group (placebo and atomoxetine) was calculated using linear mixed models in an intent-to-treat an analysis.
Time Frame: baseline and weekly through week 12 post randomization
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 35 | 35
units on a scale | 18.61 [15.13 to 22.08] | 18.19 [13.41 to 22.97]

2. Secondary Outcome: Time Line Followback Interview (TLFB)
Description: The TLFB assesses the number of days in which a substance was used in the past 28 days. The TLFB is administered by the clinician and uses a 28-day calendar with anchor points to record this information. This instrument relies on confidential self-report of the adolescent participant. The result is reported as mean change in the number of days used substances in the past 28 days from baseline to the end of treatment using linear mixed models in an intent-to-treat analysis.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 35 | 35
days | -2.24 [-5.67 to 1.18] | -5.78 [-9.21 to 2.35]

3. Secondary Outcome: Side Effect Form for Children and Adolescents (SEFCA)
Description: The SEFCA is a clinician-administered instrument that systematically assesses 52 possible side effects and rates them on a scale of 0 (not present) to 3 (severe). The instrument relies on confidential, self-report of the adolescent.The number of serious adverse events was recorded by intervention assignment.
Time Frame: weekly from randomization to 12 weeks post-randomization
Measure: Number; unit: Number of serious adverse events
Arm/Group | Placebo | Atomoxetine
Number analyzed (Participants) | 35 | 35
Number of serious adverse events | 1 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 1/35 | 1/35
Other Adverse Events (participants affected / at risk) | 16/35 | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | Atomoxetine (N=35)
suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) — One participant on placebo attempted to shoot himself with a revolver. There was no bullet in the chamber.
Overdose (Nervous system disorders) | 0 (0) | 1 (1) — One participant on atomoxetine took an overdose of bupropion tablets because he was told he could hallucinate by doing so. He had a seizure, which was treated in a local emergency room.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=35) | Atomoxetine (N=35)
difficulty concentrating (Psychiatric disorders) | 16 (16) | 23 (23) — Participants reporting difficulty with focusing.

LIMITATIONS AND CAVEATS:
1. The study was not powered to assess safety.
2. Participants received individual motivational interviewing/cognitive behavioral therapy for substance treatment. The results may not generalize to samples receiving different behavioral treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No